CLINICAL TRIAL: NCT01278862
Title: Clinical Evaluation of Lava Digital Veneer System (DVS) Crowns
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: product no longer on market
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3M ESPE CR-10-004
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Decay
Keywords: Crowns; posterior teeth; CAD CAM crowns; digital veneer system; Lava; clinical
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DVS veneer (Experimental): veneer made by CAD/CAM method
  Interventions: Device: DVS veneer
- Conventional veneer (Active Comparator): Veneer made by laboratory technician
  Interventions: Device: Conventional Veneer

INTERVENTIONS:
Device: DVS veneer — CAD/CAM milled porcelain veneer for Lava crown
  Other Names: Lava digital veneer system
  Arms: DVS veneer
Device: Conventional Veneer — CAD/CAM milled Lava crown with lab fabricated veneer
  Other Names: Lava Crown
  Arms: Conventional veneer

SUMMARY:
Study aim is to compare Lava Computer Aided Design / Computer Aided Milling Computer Aided Machining (CAD/CAM)crowns that are veneered (covered) with porcelain that has been milled using CAD/CAM, with similar CAD/CAM Lava crowns that have been veneered with a hand fabricated porcelain covering.

DETAILED DESCRIPTION:
Veneers will be randomly allocated to study crowns. Study crowns will be evaluated over three years. The test porcelain veneer is CAD/CAM milled as a veneer shell that is then fused to the CAD/CAM milled Lava crown to make the final crown to be cemented in the patient's mouth. This may be a more predictable technique in the fabrication of Lava crowns than current conventional methods.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Have at least one decayed back tooth in need of a crown
* Study tooth to be an upper or lower premolar or molar tooth/ teeth
* Study tooth to be vital and asymptomatic at start of study

Exclusion Criteria:

* Teeth which are non vital, have had root canal treatment
* Teeth which are pulp capped
* Sensitive teeth
* Significant untreated dental disease including periodontitis and rampant decay
* Pregnant or lactating women
* Patients with allergies to any of the materials to be used in the study
* Unable to attend the recall appointments

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Fasbinder, DDS, Principal Investigator — Univ of Michigan School of Dentistry
Locations (1):
- University of Michigan Dental School, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Crowns
Groups:
- Conventional Veneer: Veneer made by laboratory technician
  DVS veneer: CAD/CAM milled porcelain veneer for Lava crown
Period: Overall Study
Arm/Group | DVS Veneer | Conventional Veneer
Started (Total # of participants equaled 77; Some subjects received more than one crown (max, of 2).) | 45; 50 Crowns | 43; 50 Crowns
Completed (1 subject with one of each crown placed was lost follow-up) | 44; 49 Crowns | 42; 49 Crowns
Not Completed | 1; 1 Crowns | 1; 1 Crowns
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: 77 patients enrolled in study- Each patient received a maximum of two crowns. Consequently, the total # of participants is less than the sum of participants in each group. If more than one crown placed, crowns may have been distributed as one from each group or two of the same group.
Units Other Than Participants: Crowns
Groups:
- Total: Total of all reporting groups
Arm/Group | DVS Veneer | Conventional Veneer | Total
Number analyzed (Participants) | 45 | 43 | 77
Number analyzed (Crowns) | 50 | 50 | 100
Age, Categorical [Count of Units; unit: Crowns] — Population: Some patients received more than one crown. Such patients may have received multiple (maximum 2) of the same type of crown or a crown from both arms.
  Crowns
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 44 | 46 | 90
    >=65 years | 6 | 4 | 10
Sex: Female, Male [Count of Units; unit: Crowns] — Population: Some patients received more than one crown. Such patients may have received multiple (maximum 2) of the same type of crown or a crown from both arms.
  Crowns
    Female | 38 | 33 | 71
    Male | 12 | 17 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Performance of Crowns Via Modified United States Public Health Service (USPHS) Criteria
Description: Performance reported as the % of teeth with perfect (alpha/A) scores. USPHS criteria: Color Match ( A=Ideal, B=perceptible mismatch but acceptable, C=obvious mismatch and unacceptable); Margin Adaptation (A=no visible crevice, B=crevice along <50% margin>1mm depth, C=crevice along>50% margin >1mm depth); Margin discoloration (A=none, B=Surface stain non penetrating, C=Penetrating; Surface Finish (A=smooth, B=moderately uniformly rough, C=significant pitts/voids; Crown Fracture (A=none, B=small but repairable, C= coping exposed/complete delamination; Proximal Contact (A=firm resistance to floss/ideal contact, B=light resistance/variable breadth, C=open; Sensitivity (A=none, B= slight but not uncomfortable, C=severe; Caries (A=no evidence, B= evident but repairable, C=evident/not repairable.
Time Frame: 1 year
Population: Number of crowns evaluated within each group after 1 year in vivo
Measure: Count of Units; unit: Crowns
Units Other Than Participants: Crowns
Arm/Group | DVS Veneer | Conventional Veneer
Number analyzed (Participants) | 44 | 42
Number analyzed (Crowns) | 49 | 49
Crowns
  Color Match | 49 | 46
  Margin Adaptation | 49 | 49
  Margin Discoloration | 49 | 48
  Surface Finish | 49 | 49
  Caries | 49 | 49
  Crown Fracture | 48 | 48
  Sensitivity | 49 | 49
  Proximal Contact - Mesial | 48 | 47
  Proximal Contace - Distal: number analyzed (Crowns) | 43 | 42
  Proximal Contace - Distal | 42 | 41
Statistical Analysis 1: Comparison: DVS Veneer vs Conventional Veneer; null hypothesis no difference in color match; Test type: Superiority or Other; p = 0.2423, Fisher Exact
Statistical Analysis 2: Comparison: DVS Veneer vs Conventional Veneer; null hypothesis no difference in margin discoloration; Test type: Superiority; p > 0.999, Fisher Exact
Statistical Analysis 3: Comparison: DVS Veneer vs Conventional Veneer; null hypothesis no difference in crown fracture; Test type: Superiority; p > 0.999, Fisher Exact
Statistical Analysis 4: Comparison: DVS Veneer vs Conventional Veneer; Null hypothesis no difference in Proximal Contact - Mesial; Test type: Superiority or Other; p > 0.999, Fisher Exact
Statistical Analysis 5: Comparison: DVS Veneer vs Conventional Veneer; Null hypothesis no difference in proximal contact - distal; Test type: Superiority or Other; p > 0.999, Fisher Exact

2. Primary Outcome: Gingival/Periodontal Health Based on Loe & Stillness Index, 1963.
Description: Performance reported as the # of crowns exhibiting 0, 1, 2 and 3 index score. Gingival Index (0=normal, 1=mild inflammation, 2=moderate inflammation, 3=severe inflammation. Plaque Index (0= none, 1= observed only via probe at on tooth surface at gingival crest, 2=moderate accumulation along gingival margin and adjacent tooth, 3= abundant plaque along gingival margin and adjacent tooth.
Time Frame: 1 year
Population: Number of crowns evaluated within each group after 1 year in vivo
Measure: Number; unit: Crowns
Units Other Than Participants: Crowns
Arm/Group | DVS Veneer | Conventional Veneer
Number analyzed (Participants) | 44 | 42
Number analyzed (Crowns) | 49 | 49
Crowns
  Gingival Index=0 | 49 | 48
  Gingival Index=1 | 0 | 1
  Plaque Index=0 | 42 | 45
  Plaque Index=1 | 7 | 4
Statistical Analysis 1: Comparison: DVS Veneer vs Conventional Veneer; null hypothesis no difference in gingival index; Test type: Superiority; p > 0.999, Fisher Exact
Statistical Analysis 2: Comparison: DVS Veneer vs Conventional Veneer; null hypothesis no difference in plaque index; Test type: Superiority; p = 0.5240, Fisher Exact

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | DVS Veneer | Conventional Veneer
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/43
Other Adverse Events (participants affected / at risk) | 0/45 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No